CLINICAL TRIAL: NCT00121121
Title: A Phase Ib Vaccine Trial Evaluating the Safety and Immunogenicity of HIV Lipopeptides by Two Administration Routes (Intramuscular And Intradermal) in Healthy Adult Volunteers. ANRS VAC16 Trial
Brief Title: Safety of Intradermal Versus Intramuscular Administration of HIV Lipopeptides in HIV Uninfected Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS VAC16
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2005-11

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: HIV Vaccines; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: Lipopeptides LIPO-4

SUMMARY:
Intramuscular (IM) administration of HIV lipopeptide vaccines have been shown to be able to induce HIV-1-specific T cell-mediated immune responses. The objective of this trial was to evaluate the safety and immunogenicity of LIPO-4 vaccine (HIV lipopeptides including 4 peptides from Gag, Pol, RT and Nef HIV-1 proteins, each peptide linked to TT) intradermally (ID) compared to IM administration.

DETAILED DESCRIPTION:
Dose-sparing strategies that use intradermal (ID) delivery of vaccines may be one approach for improving a vaccines immunogenicity and reducing the cost of vaccines.

In this study, 68 HIV-negative healthy adult volunteers, 21-55 years old, all belonging to the "Volunteers for a Vaccine" network set up by ANRS, were randomized to receive at weeks 0, 4, and 12, either 3 IM doses of 0.5 ml of LIPO-4 containing 500 µg of each peptide (n= 35 volunteers), or 3 ID doses of 0.1 ml, containing 100 µg of each peptide (n=33 volunteers). Total follow-up was 48 weeks. Safety was assessed clinically and by laboratory tests. Participants were given diary cards to record adverse events. HIV-1 immune responses were assessed by ELISPOT and lymphoproliferative assay at weeks 0, 2, 6, 14, 24, and 48

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected
* Acceptable methods of contraception for females of reproductive potential
* Good general health
* Signed written inform consent

Exclusion Criteria:

* Risk to be infected by HIV virus
* Uveitis, chronic lyme disease, active syphilis, active mycobacterial diseases or sarcoidosis
* Autoimmune disease or immunodeficiency
* Medical history of food allergy, Lyell's or Steven Johnson's disease, unstable asthma
* Active, generalized eczema or chronic urticaria
* Blood products within 2 months prior to first study vaccine administration
* HIV vaccines in prior HIV vaccine trial or participation in an immunomodulator study
* Vaccines within 30 days prior to first study vaccine administration
* Pregnant
* Long-term immunosuppressive or immunomodulator medications or within 6 months to first study vaccine administration
* Blood transfusion within 6 months to first study vaccine administration
* Treated with extracted pituitary hormones

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70
Dates: Start 2004-07; Study Completion 2005-12

PRIMARY OUTCOMES:
Clinical and biological safety (over or equal to degree two of a adverse event grading scale) of LIPO-4 by ID and IM routes during the study

SECONDARY OUTCOMES:
Comparaison of CD4 positive cells responses using
lymphoprolifération test and CD8 positive cells responses using the capacity of these cells to synthesize IFN following stimulation with peptides of interest (ELISPOT IFN test) following IM or ID administration at weeks 2, 6, 14, 24, and 48

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, MD, Principal Investigator — Hopital Cochin Paris, Centre Cochin-Pasteur d'essais vaccinaux; Christine Durier, MD, Study Director — Inserm SC10
Locations (1):
- Hopital Cochin Centre Cochin-Pasteur d'Essais vaccinaux, Paris, France

REFERENCES:
- [Derived] Launay O, Durier C, Desaint C, Silbermann B, Jackson A, Pialoux G, Bonnet B, Poizot-Martin I, Gonzalez-Canali G, Cuzin L, Figuereido S, Surenaud M, Ben Hamouda N, Gahery H, Choppin J, Salmon D, Guerin C, Bourgault Villada I, Guillet JG; ANRS VAC16 Study Group. Cellular immune responses induced with dose-sparing intradermal administration of HIV vaccine to HIV-uninfected volunteers in the ANRS VAC16 trial. PLoS One. 2007 Aug 22;2(8):e725. doi: 10.1371/journal.pone.0000725. PMID 17712402